CLINICAL TRIAL: NCT06368661
Title: Dietary Factors Associated to Colorectal Premalignant Lesions (COLOMAR-1)
Status: Recruiting | Type: Observational
Sponsor: Fundación Vithas (Other)
Collaborators: CEU San Pablo University (Other)
Responsible Party: Sponsor
Other Study IDs: 23.79 Colo-MAR 1
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-04

CONDITIONS: Nutrition Related Neoplasm/Cancer
Keywords: Fish; Colon cancer; Rectal cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Colon mucosa and blood samples will be taken to find alkylating signature and dismiss other genetic patterns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to find a correlation between fish protein intake and other dietary habits and colorectal premalignant lesions in healthy volunteers. It also aims to describe gut microbial profiles for each dietary pattern, in order to elucidate the role of fish intake in cancer prevention.

DETAILED DESCRIPTION:
Colorectal cancer incidence is increasing in developed countries specially among young adults due to risk factors as modern dietary, smoking, low physical exercise and obesity. Some foods (fruits, vegetables, nuts, other seeds and legumes) are assumed to prevent occurrence of colorectal cancer, while red and processed meat intake are strongly associated with increased risk of colorectal tumors. However, evidence on fish intake is still scarce, and the mechanisms and drivers of their potential health benefits are also only partially known. On the other hand, colonoscopy remains the gold standard for colon cancer screening. Our study aims to explore the relationship among fish intake, microbiota and molecular alterations during a colonoscopy screening program of healthy volunteers. This is a preliminary proof-of-concept study (ColoMAR-1) to evaluate the feasibility of the entire research program (ColoMAR-2).

The main objectives of this pilot are:

1. To determinate the feasibility of the entire research project obtaining data for all the study participants (colonoscopy, blood sample, feces sample and dietary questionnaire).
2. To evaluate the presence of precancerous lesions (colonic polyps) and colorectal malignant tumors in all the participants.
3. To find molecular alterations (Alkylating signature) in normal mucosa of right and left-sided colon samples.
4. To describe microbiota composition in all the participants.
5. To determinate correlation between dietary habits and clinical and molecular findings of the study.
6. To calculate the overall sample size of the entire research program (ColoMAR-2) in base to dietary patterns and Alkylating signature prevalence of the participants)

ELIGIBILITY:
Inclusion Criteria:

* 45 years old or more.
* Be willing to participate in the study.

Exclusion Criteria:

* Pregnancy
* Previous colorectal cancer.
* Familial colorectal cancer syndrome.
* Previous colonoscopy and colon polypectomy (last five years ).
* Inflammatory bowel disease.
* Medical contraindication for colonoscopy at investigator´s criteria.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers from the general population above 45 years old.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dietary habits registry from participants: the dietary intake | Dietary habits will be taken by an online specific Food Frequency Questionnaire (FFQ) for Spanish population. The data analysis will be taken at baseline outcome. 3 months
  Dietary habits will be taken by an online specific Food Frequency Questionnaire (FFQ) for Spanish population. The data analysis will be taken at baseline outcome.
Biomarkers in colon mucosa, precancerous lesions and colorectal cancer | 3 months
  Alkylating signature will be determined in normal mucosa of right and left colon, premalignant lesions and colorectal cancer
Gut microbiota profile | 4 months
  Differences in profile of gut microbiota among participants with and without precancerous lesions and colorectal cancer will be evaluated. Differences in profile of gut microbiota among different profiles of dietary habits will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ciro Cabezas Checchi, Vigo, Pontevedra, Spain